CLINICAL TRIAL: NCT05964725
Title: The Study on Effect and Neural Network Mechanism of Transcranial Direct Current Stimulation for Sudden Deafness With Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSKY-2022-499-02
Record Dates: First submitted 2023-07-16; First posted 2023-07-28 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Tinnitus, Subjective; Sudden Deafness; Transcranial Direct Current Stimulation; Double-Blind Method; Female; Male; Human; Treatment Outcome
Keywords: Acute subjective tinnitus; Clinical trial; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Tinnitus; Hearing Loss, Sudden | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants in the included studies were randomized 1:1 by statisticians. The statistician will number the subjects using a computer-generated random number table, then arrange them in order of number size, and then randomly divide the subjects into random blocks of length 2 or 4 to complete the randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the whole clinical research process, the subjects and researchers participating in the efficacy and safety evaluation should be in a blind state, that is, neither of them knows the specific intervention measures given to the subjects. For participant, the treatment equipment is exactly the same between the two groups. Also, 10 seconds sham stimulation at the beginning of treatment is set in the control group for minimizing risk of participants being able to guess treatment allocation. The randomized allocation is completed by a unified randomization center. Therefore, the investigators in each center just know "A" or "B" for the allocation information of each participant. For outcomes assessors, they are only responsible for baseline and follow-up assessment during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receive traditional medical therapy and transcranial direct current stimulation (Experimental): intravenous methylprednisolone infusion (dose of 1 mg/kg/day, maximum 60 mg/day) for 5 to 10 days. Patients included in this study were routinely examined and tested for audiometry, including otoscopy, pure tone audiometry, acoustic impedance, brainstem evoked potential, and tinnitus detection. After completion, the 32-guide EEG collector from Bricon was used to collect changes in neural activity in all subjects.
  Interventions: Device: Receive traditional medical therapy and transcranial direct current stimulation
- Receive traditional medical therapy and sham stimulation (Sham Comparator): Similarly, intravenous methylprednisolone infusion (dose of 1 mg/kg/day, maximum 60 mg/day) for 5 to 10 days. By controlling the tDCS stimulator to mimic only the first 30 seconds of tDCS stimulation, after 30 seconds of pathway resistance control, so that the stimulation intensity is below the threshold, without giving real stimulation, in this process, the position of the stimulation target is not changed, and the rest of the operation is the same.
  Interventions: Device: Receive traditional medical therapy and sham stimulation

INTERVENTIONS:
Device: Receive traditional medical therapy and transcranial direct current stimulation — Equipment used: Bricon tDCS stimulator, high-precision electrode stimulation method Stimulant dose: 1.5mA Stimulation time: 20 minutes/time, continuous treatment for 5 days Stimulation course: 5 days/course Stimulation target: left auditory cortex area, i.e., under system 10-20, left T3 position.
  Arms: Receive traditional medical therapy and transcranial direct current stimulation
Device: Receive traditional medical therapy and sham stimulation — By controlling the tDCS stimulator to mimic only the first 30 seconds of tDCS stimulation, after 30 seconds of pathway resistance control, so that the stimulation intensity is below the threshold, without giving real stimulation, in this process, the position of the stimulation target is not changed, and the rest of the operation is the same.
  Arms: Receive traditional medical therapy and sham stimulation

SUMMARY:
This clinical study is prospective, single-center, randomized, controlled, double-blind clinical trail, which entitled transcranial electrical stimulation for the treatment of acute tinnitus approved by Sun Yat-sen University, and intends to recruit 86 patients with sudden deafness and tinnitus. For acute subjective tinnitus, a common otological disease, the study gave the experimental group patients received tDCS with electrodes positioned over the left temporal cortex for 5 days. To assess the efficacy of conventional medical therapy and tDCS by comparing changes in anterior and posterior tinnitus-related subjective scale scores, such as THI, VAS, BAI, BDI, PSQI, and hearing recovery, in patients who received tDCS, to determine whether tDCS is effective in improving acute tinnitus, and whether it is superior to conventional tinnitus treatment. In addition, the study will continue to follow patients for 1 month,3 months, and 6 months after the end of treatment to observe the long-term sustained efficacy of tDCS. This clinical trail will also evaluate tDCS from the perspective of compliance and safety, and explore the factors affecting the efficacy of this therapy.

DETAILED DESCRIPTION:
Sample size estimation:

On-site recruitment will be conducted in the otolaryngology clinic for eligible patients with sudden deafness and tinnitus, with dedicated personnel to recruit subjects, with a total of at least 86 expected recruitment. In order to retain subjects, staff will tell them about the benefits of inclusion in clinical studies for sudden deafness with tinnitus, and actively add subjects' contact information to provide relevant consulting services for subjects during clinical studies. During follow-up, participants will be provided with a free tinnitus-related assessment test to motivate.

Plan for missing data： Screening failure, i.e. subjects did not meet the inclusion and exclusion criteria, or subjects withdrew informed consent, among other things for reasons why it was not included in this clinical study. Study subjects who failed to screen will be pressed according to their own condition Provide appropriate treatment according to clinical guidelines. This subset of subjects will not be included in clinical studies.

Statistical analysis plan:

When considering the influence of baseline, the continuous variables were analyzed by covariance analysis, and the qualitative indicators were tested by CMH test or logistic regression.

Primary analysis： Using covariance analysis to compare the different changes of THI scores between two groups after 5 days treatment, controlled for age and baseline THI.

Secondary analysis： Using covariance analysis to compare the different changes of VAS, BAI, BDI, PSQI scores between two groups after 5 days treatment, controlled for age and baseline values corresponding to each scale.

Using a repeated measure ANOVA to compare the different changes of THI, VAS, BAI, BDI, PSQI between two groups at 1, 3 and 6 follow-up visits.

Using Chi square test or Fisher exact test to compare the different efficient rate between two groups after 5 days treatment.

Exploratory analysis:

Using multiple linear regression analysis to explore the factors affecting the short-term and long -term efficacy of the two treatments, such as age, hearing loss threshold, tinnitus loudness, tinnitus frequency and so on.

Using Independent two sample t-test or nonparametric analysis to compare the differences in EEG- or fMRI-related indicators between two groups.

Safety analysis:

Using Pearson's chi-square test to compare the difference of adverse event incidence rate between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tinnitus as the main complaint: patients subjectively feel sound in the ear or deep part of the head without internal or external sound stimulation, with or without hearing loss, and seek medical treatment
* Patients with sudden deafness with tinnitus whose course is less than 1 month and have not received any drug treatment
* Age 18-60 years
* Tinnitus frequency is 125-8000 Hz

Exclusion Criteria:

* Patients with conductive deafness, history of middle ear surgery, pulsatile tinnitus caused by vascular aberration and tinnitus cause by Meniere disease
* History of head trauma, central nervous system disease, mental disease, and drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-11-23 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Tinnitus Handicap Inventory (THI) scores for short-term efficacy assessment | From baseline to after 5 days treatment
  Difference in the change of THI scores between two groups after 5 days treatment. The THI evaluates the severity of tinnitus in terms of emotion and function. The global scores of THI range from 0 (no disability) to 100 (serve disability).

SECONDARY OUTCOMES:
Changes in scores of Visual Analog Scale (VAS) for short-term efficacy assessment | From baseline to after 5 days treatment
  Difference in the change of VAS scores between two groups after 5 days treatment. The total VAS scores range from 0 (negligible) to 10 (too noisy to tolerate), reflecting the loudness of tinnitus patients feel.
Changes in scores of Beck Anxiety Inventory (BAI) for short-term efficacy assessment | From baseline to after 5 days treatment
  Difference in the change of BAI scores between two groups after 5 days treatment. The total BAI scores range from 0 (normal) to 63 (serve anxiety), reflecting the degree of anxiety.
Changes in scores of Beck Depression Inventory (BDI) for short-term efficacy assessment | From baseline to after 5 days treatment
  Difference in the change of BDI scores between two groups after 5 days treatment. The total BDI scores range from 0 (normal) to 63 (serve depression), reflecting the degree of depression.
Changes in scores of Pittsburgh sleep quality index (PSQI) for short-term efficacy assessment | From baseline to after 5 days treatment
  Difference in the change of PSQI scores between two groups after 5 days treatment. The total PSQI scores range from 0 (sleep well) to 21 (quite poor sleep), reflecting the sleep quality.
Changes of Tinnitus Handicap Inventory (THI) scores in the two groups for long-term efficacy assessment | From 1-month follow-up visit to 6-month follow-up visit
  Difference in changes of THI between two groups from 1-month follow-up visit to 6-month follow-up visit. The THI evaluates the severity of tinnitus in terms of emotion and function. The global scores of THI range from 0 (no disability) to 100 (serve disability).
Changes of Visual Analog Scale (VAS) scores in the two groups for long-term efficacy assessment | From 1-month follow-up visit to 6-month follow-up visit
  Difference in changes of VAS between two groups from 1-month follow-up visit to 6-month follow-up visit. The total VAS scores range from 0 (negligible) to 10 (too noisy to tolerate), reflecting the loudness of tinnitus patients feel.
Changes of Beck Anxiety Inventory (BAI) scores in the two groups for long-term efficacy assessment | From 1-month follow-up visit to 6-month follow-up visit
  Difference in changes of BAI between two groups from 1-month follow-up visit to 6-month follow-up visit. The total BAI scores range from 0 (normal) to 63 (serve anxiety), reflecting the degree of anxiety.
Changes of Beck Depression Inventory (BDI) scores in the two groups for long-term efficacy assessment | From 1-month follow-up visit to 6-month follow-up visit
  Difference in changes of PSQI between two groups from 1-month follow-up visit to 6-month follow-up visit. The total BDI scores range from 0 (normal) to 63 (serve depression), reflecting the degree of depression.
Changes of Pittsburgh sleep quality index (PSQI) scores in the two groups for long-term efficacy assessment | From 1-month follow-up visit to 6-month follow-up visit
  Difference in changes of PSQI between two groups from 1-month follow-up visit to 6-month follow-up visit. The total PSQI scores range from 0 (sleep well) to 21 (quite poor sleep), reflecting the sleep quality.
The effective rate of relieving sudden deafness with tinnitus in the two groups | From baseline to after 5 days treatment
  Group effective rate = number of patients in each group who completed 5 days of treatment and whose THI score decreased by ≥ 7 points / number of patients in each group who completed 5 days of treatment.
The difference of functional connectivity based on resting state electroencephalogram (EEG) between the two groups | From 1-month follow-up visit to 6-month follow-up visit
  The difference of functional connectivity based on resting state electroencephalogram (EEG) in the two groups from 1-month follow-up visit to 6-month follow-up visit. The functional connectivity is defined as the correlation between two different brain regions based on coherence or phase synchronization.
The difference of effective connectivity based on resting state electroencephalogram (EEG) between the two groups | From 1-month follow-up visit to 6-month follow-up visit
  The difference of effective connectivity based on resting state electroencephalogram (EEG) in the two groups from 1-month follow-up visit to 6-month follow-up visit. The effective connectivity is defined as the directed functional connectivity between two brain regions based on granger causality analysis.
The difference of functional connectivity based on functional magnetic resonance imaging (fMRI) between the two groups | From 1-month follow-up visit to 6-month follow-up visit
  The difference of functional connectivity based on functional magnetic resonance imaging (fMRI) in the two groups from 1-month follow-up visit to 6-month follow-up visit. The functional connectivity is defined as the Pearson's correlation between two different brain regions.
The difference of effective connectivity based on functional magnetic resonance imaging (fMRI) between the two groups | From 1-month follow-up visit to 6-month follow-up visit
  The difference of effective connectivity based on functional magnetic resonance imaging (fMRI) in the two groups from 1-month follow-up visit to 6-month follow-up visit. The effective connectivity is defined as the directed functional connectivity between two brain regions based on granger causality analysis.

OTHER OUTCOMES:
Incidence of treatment-related adverse events | From baseline to 6-month follow-up visit
  Treatment related adverse events in two groups include: auditory system related adverse reactions caused by treatment, such as auricle burn, earache, hearing loss, tinnitus aggravation, and head injury Dizziness, headache, palpitation, vomiting and other non auditory system related adverse reactions. Incidence of adverse events = number of treatment-related adverse events during treatment / total number of participants in treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yuexin Cai, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chandrasekhar SS, Tsai Do BS, Schwartz SR, Bontempo LJ, Faucett EA, Finestone SA, Hollingsworth DB, Kelley DM, Kmucha ST, Moonis G, Poling GL, Roberts JK, Stachler RJ, Zeitler DM, Corrigan MD, Nnacheta LC, Satterfield L. Clinical Practice Guideline: Sudden Hearing Loss (Update). Otolaryngol Head Neck Surg. 2019 Aug;161(1_suppl):S1-S45. doi: 10.1177/0194599819859885. PMID 31369359
- [Background] Rah YC, Park KT, Yi YJ, Seok J, Kang SI, Kim YH. Successful treatment of sudden sensorineural hearing loss assures improvement of accompanying tinnitus. Laryngoscope. 2015 Jun;125(6):1433-7. doi: 10.1002/lary.25074. Epub 2014 Dec 4. PMID 25476777
- [Background] Klemm E, Bepperling F, Burschka MA, Mosges R; Study Group. Hemodilution therapy with hydroxyethyl starch solution (130/0.4) in unilateral idiopathic sudden sensorineural hearing loss: a dose-finding, double-blind, placebo-controlled, international multicenter trial with 210 patients. Otol Neurotol. 2007 Feb;28(2):157-70. doi: 10.1097/01.mao.0000231502.54157.ad. PMID 17255882
- [Background] Westerlaken BO, de Kleine E, van der Laan B, Albers F. The treatment of idiopathic sudden sensorineural hearing loss using pulse therapy: a prospective, randomized, double-blind clinical trial. Laryngoscope. 2007 Apr;117(4):684-90. doi: 10.1097/mlg.0b013e3180316d3b. PMID 17415139
- [Background] Zhou GP, Chen YC, Li WW, Wei HL, Yu YS, Zhou QQ, Yin X, Tao YJ, Zhang H. Aberrant functional and effective connectivity of the frontostriatal network in unilateral acute tinnitus patients with hearing loss. Brain Imaging Behav. 2022 Feb;16(1):151-160. doi: 10.1007/s11682-021-00486-9. Epub 2021 Jul 23. PMID 34296381
- [Background] Aldhafeeri FM, Mackenzie I, Kay T, Alghamdi J, Sluming V. Neuroanatomical correlates of tinnitus revealed by cortical thickness analysis and diffusion tensor imaging. Neuroradiology. 2012 Aug;54(8):883-92. doi: 10.1007/s00234-012-1044-6. Epub 2012 May 22. PMID 22614806
- [Background] Cai Y, Xie M, Su Y, Tong Z, Wu X, Xu W, Li J, Zhao F, Dang C, Chen G, Lan L, Shen J, Zheng Y. Aberrant Functional and Causal Connectivity in Acute Tinnitus With Sensorineural Hearing Loss. Front Neurosci. 2020 Jun 30;14:592. doi: 10.3389/fnins.2020.00592. eCollection 2020. PMID 32714128
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Teismann H, Wollbrink A, Okamoto H, Schlaug G, Rudack C, Pantev C. Combining transcranial direct current stimulation and tailor-made notched music training to decrease tinnitus-related distress--a pilot study. PLoS One. 2014 Feb 25;9(2):e89904. doi: 10.1371/journal.pone.0089904. eCollection 2014. PMID 24587113
- [Background] Pal N, Maire R, Stephan MA, Herrmann FR, Benninger DH. Transcranial Direct Current Stimulation for the Treatment of Chronic Tinnitus: A Randomized Controlled Study. Brain Stimul. 2015 Nov-Dec;8(6):1101-7. doi: 10.1016/j.brs.2015.06.014. Epub 2015 Jun 27. PMID 26198363
- [Background] Vanneste S, De Ridder D. Bifrontal transcranial direct current stimulation modulates tinnitus intensity and tinnitus-distress-related brain activity. Eur J Neurosci. 2011 Aug;34(4):605-14. doi: 10.1111/j.1460-9568.2011.07778.x. Epub 2011 Jul 25. PMID 21790807
- [Background] Vanneste S, Plazier M, Ost J, van der Loo E, Van de Heyning P, De Ridder D. Bilateral dorsolateral prefrontal cortex modulation for tinnitus by transcranial direct current stimulation: a preliminary clinical study. Exp Brain Res. 2010 May;202(4):779-85. doi: 10.1007/s00221-010-2183-9. Epub 2010 Feb 26. PMID 20186404
- [Background] Vanneste S, Focquaert F, Van de Heyning P, De Ridder D. Different resting state brain activity and functional connectivity in patients who respond and not respond to bifrontal tDCS for tinnitus suppression. Exp Brain Res. 2011 Apr;210(2):217-27. doi: 10.1007/s00221-011-2617-z. Epub 2011 Mar 25. PMID 21437634
- [Background] Faber M, Vanneste S, Fregni F, De Ridder D. Top down prefrontal affective modulation of tinnitus with multiple sessions of tDCS of dorsolateral prefrontal cortex. Brain Stimul. 2012 Oct;5(4):492-8. doi: 10.1016/j.brs.2011.09.003. Epub 2011 Oct 5. PMID 22019079
- [Background] Frank E, Schecklmann M, Landgrebe M, Burger J, Kreuzer P, Poeppl TB, Kleinjung T, Hajak G, Langguth B. Treatment of chronic tinnitus with repeated sessions of prefrontal transcranial direct current stimulation: outcomes from an open-label pilot study. J Neurol. 2012 Feb;259(2):327-33. doi: 10.1007/s00415-011-6189-4. Epub 2011 Aug 2. PMID 21808984
- [Background] Vanneste S, Langguth B, De Ridder D. Do tDCS and TMS influence tinnitus transiently via a direct cortical and indirect somatosensory modulating effect? A combined TMS-tDCS and TENS study. Brain Stimul. 2011 Oct;4(4):242-52. doi: 10.1016/j.brs.2010.12.001. Epub 2011 Jan 1. PMID 22032739
- [Background] Yakunina N, Nam EC. Direct and Transcutaneous Vagus Nerve Stimulation for Treatment of Tinnitus: A Scoping Review. Front Neurosci. 2021 May 28;15:680590. doi: 10.3389/fnins.2021.680590. eCollection 2021. PMID 34122002
- [Background] Gordon PC, Zrenner C, Desideri D, Belardinelli P, Zrenner B, Brunoni AR, Ziemann U. Modulation of cortical responses by transcranial direct current stimulation of dorsolateral prefrontal cortex: A resting-state EEG and TMS-EEG study. Brain Stimul. 2018 Sep-Oct;11(5):1024-1032. doi: 10.1016/j.brs.2018.06.004. Epub 2018 Jun 18. PMID 29921529
- [Background] Joos K, De Ridder D, Van de Heyning P, Vanneste S. Polarity specific suppression effects of transcranial direct current stimulation for tinnitus. Neural Plast. 2014;2014:930860. doi: 10.1155/2014/930860. Epub 2014 Apr 10. PMID 24812586